CLINICAL TRIAL: NCT04107909
Title: Three-port Versus Four-port Laparoscopic Cholecystectomy: A Prospective Comparative Study
Brief Title: Laparoscopic Cholecystectomy:
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Abdelfatah Elshreef, general surgery, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: lapgb
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 ports (Other): 3port operation
  Interventions: Procedure: laparoscopic cholecystectomy
- 4 port (Other): 4 port operation
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — Both four port and three port LC is performed With the patient in supine position, with the surgeon and assistant on the left side and the monitor on the right side. Head up and right up position is employed during surgery in both the groups. Pneumoperitoneum of 12mmHg is created using open Hassan's method through the umbilical port.
  In 3 port a 5.5 mm umbilical visiport for 5 mm lens 30 degree A second 10 mm trocar is placed inferior to the sternum at the midline, while the third 5mm trocar is placed 4-5cm inferior to the right costal margin on the right midclavicular line. For the four port LC, additional 5mm port is placed in the sub costal region at the anterior axillary line. Posterior dissection and delineation of The Calot's triangle is done. Then, the cystic artery and cystic duct are identified, isolated, doubly clipped and divided. The gallbladder is removed through the umbilical port using a 10mm gallbladder extractor.

SUMMARY:
Various modifications have been tried in laparoscopic cholecystectomy since its introduction. One, two and three port LC have been performed on limited scale. we aim to compare three port LC with four port LC in patients with cholelithiasis. The main objective of this study is to evaluate the outcome of 3 ports LC for treatment of cholelithiasis by comparing the result with 4 ports LC with respect to safety and efficacy.

DETAILED DESCRIPTION:
Various modifications have been tried in laparoscopic cholecystectomy since its introduction. One, two and three port LC have been performed on limited scale. we aim was to compare three port LC with four port LC in patients with cholelithiasis. The main objective of this study was to evaluate the outcome of 3 ports LC for treatment of cholelithiasis by comparing the result with 4 To study the efficacy and feasibility of 3 port and 4 port lap cholecystetctomy.

1. To compare the intraoperative and post-operative complications of 3 port and 4 port lap cholecystectomy

1. Operative time,
2. Days of hospital stay.
3. complication
4. post-operative pain ports LC with respect to safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patient between 25 and 65 years
2. Diagnosis of chronic cholecystitis, symptomatic cholelithiasis

Exclusion Criteria:

1. Choledocholithiasis
2. Severe Acute Calculus Pancreatitis
3. Severe co-morbid conditions (uncontrolled diabetes, Hypertension, severe direct hyper bilirubinemia) 4 . Previous operation or adhesion

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
compare between the prognosis of three port and four port laproscpic cholecyctectomy | 3 years

REFERENCES:
- [Background] Muhe E. [Laparoscopic cholecystectomy--late results]. Langenbecks Arch Chir Suppl Kongressbd. 1991:416-23. doi: 10.1007/978-3-642-95662-1_189. German. PMID 1838946
- [Background] Traverso LW. Carl Langenbuch and the first cholecystectomy. Am J Surg. 1976 Jul;132(1):81-2. doi: 10.1016/0002-9610(76)90295-6. PMID 782269
- [Background] Trichak S. Three-port vs standard four-port laparoscopic cholecystectomy. Surg Endosc. 2003 Sep;17(9):1434-6. doi: 10.1007/s00464-002-8713-1. Epub 2003 Jun 13. PMID 12799892